CLINICAL TRIAL: NCT07123987
Title: Transcutaneous Auricular Vagus Nerve Stimulation on Post-Herpetic Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Hosny Ismail Easa (Other)
Responsible Party: Sponsor-Investigator, Mohamed Hosny Ismail Easa, Principal Investigator, MSc Candidate, Faculty of Physical Therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005412
Record Dates: First submitted 2025-08-12; First posted 2025-08-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Post Herpetic Neuralgia (PHN)
Keywords: Post-Herpetic Neuralgia; Neuropathic Pain; Herpes Zoster; Transcutaneous Auricular Vagus Nerve Stimulation (taVNS); Non-invasive Neuromodulation; Chronic Pain Management; Pain Relief; Randomized Controlled Trial
MeSH Terms: conditions — Neuralgia, Postherpetic; Neuralgia; Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Thirty-four male and female patients diagnosed with PHN, aged between 35 and 65 years, will be randomly allocated into two equal groups, each containing 17 patients:
  Group (A): Study group - This group will receive taVNS in addition to traditional medical treatment.
  Group (B): Control group - This group will receive the same traditional medical treatment only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): Study group (Experimental): this group will receive taVNS in addition to traditional medical treatment
  Interventions: Device: transcutaneous auricular vagus nerve stimulation (taVNS)
- Group (B): Control group (Active Comparator): this group will receive the same traditional medical treatment only
  Interventions: Other: traditional medical treatment for PHN

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation (taVNS) — Use of the EV-906 device with TENS ear clips for transcutaneous auricular vagus nerve stimulation (taVNS), applied according to the study protocol, in addition to standard medical treatment for post-herpetic neuralgia. This device meets ISO 13485, FDA QSR, and CE standards
  Arms: Group (A): Study group
Other: traditional medical treatment for PHN — Standard medical treatment for post-herpetic neuralgia as per current clinical guidelines, without the application of taVNS device.
  Arms: Group (B): Control group

SUMMARY:
The purpose of this study is to evaluate the therapeutic efficacy of transcutaneous auricular vagus nerve stimulation (taVNS) in the treatment of patients with post-herpetic neuralgia (PHN). Participants will receive taVNS in addition to standard care. The study aims to determine whether taVNS can provide significant pain relief and improve quality of life in PHN patients.

DETAILED DESCRIPTION:
Post-herpetic neuralgia (PHN) is a chronic neuropathic pain condition that persists for months or years following the resolution of herpes zoster (HZ) infection. It is characterized by persistent burning, stabbing, or shooting pain, often accompanied by allodynia and hyperalgesia, which can significantly impair quality of life. Current treatment options for PHN, including pharmacological therapies, often provide incomplete pain relief and are associated with side effects, creating a need for novel, non-invasive interventions.

This randomized controlled trial aims to evaluate the therapeutic efficacy of transcutaneous auricular vagus nerve stimulation (taVNS) as an adjunct to standard medical treatment for patients with PHN. The vagus nerve plays a crucial role in modulating pain perception and inflammatory processes, and its non-invasive stimulation through the auricular branch has shown promising analgesic effects in various chronic pain syndromes.

A total of 34 male and female participants, aged 35-65 years, diagnosed with PHN will be randomly allocated into two equal groups (17 participants per group). Group A (Experimental) will receive taVNS in addition to conventional pharmacological management, while Group B (Control) will receive conventional pharmacological management alone. The taVNS intervention will be delivered using the EV-906 device with TENS ear clips, applied according to the study protocol and safety standards (ISO 13485, FDA QSR, and CE compliance).

Pain intensity and quality will be assessed at baseline, after two weeks, and after four weeks using validated outcome measures: the Brief Pain Inventory (BPI) short form and the Short-form McGill Pain Questionnaire-2 (SF-MPQ-2). The primary outcome is the change in pain severity scores, and the secondary outcome is the change in pain interference with daily activities.

The results of this study will provide evidence regarding the clinical utility of taVNS as a safe, non-invasive, and effective adjunct therapy for PHN, with the potential to improve patient outcomes and quality of life

ELIGIBILITY:
Inclusion Criteria:

Adults aged 35-65 years diagnosed with PHN. Persistent pain for at least 3 months after herpes zoster infection. Only patients who sign the informed consent form will be included.

Exclusion Criteria:

Contraindications to taVNS such as:

1. pregnancy;
2. active implants (e.g., pacemakers, cochlear implants) or brain shunts;
3. previous neurological or psychiatric diagnoses;
4. history of addiction or substance abuse;
5. history of trauma and/or brain surgery;
6. cardiac disease;
7. acute or chronic use of medications and/or illicit drugs;
8. susceptibility to headaches and seizures. Severe cognitive impairment. Other chronic pain conditions.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory - Short Form (BPI-SF) | Administered three times: before the first treatment session, after 2 weeks, and after 4 weeks. Administration mode: Interview-based.
  the Brief Pain Inventory-Short Form (BPI SF) is a valuable tool for assessing pain severity and its impact on daily functioning on a 0-10 numeric rating scale, with higher scores indicating more severe pain.

SECONDARY OUTCOMES:
Short form McGill pain questionnaire 2 (SF-MPQ-2) | Administered three times: before the first treatment session, after 2 weeks, and after 4 weeks. Administration mode: Interview-based.
  The SF-MPQ-2 is a validated tool assessing sensory, affective, and evaluative qualities of pain. Participants rate the intensity of their pain using a 0-10 scale:
  0: No pain 10: Worst pain imaginable Participants select the rating that best reflects their experience during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa Hussein Borhan, PhD, Study Chair — Professor of Physical Therapy for Surgery Department, Faculty of Physical Therapy, Cairo University; Rofaida El Sayed El Naggar, MD, Study Director — Lecturer of Dermatology, Kasr Alainy, Faculty of Medicine, Cairo University; Doaa Atef Aly, PhD, Study Director — Lecturer of Physical Therapy for Surgery Department, Faculty of Physical Therapy, Cairo University
Locations (1):
- Faculty of Physical Therapy - Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Data will not be shared due to participant confidentiality and restrictions imposed by the institutional ethics committee